CLINICAL TRIAL: NCT05974020
Title: Investigation of the Effect of Foot Intrinsic Muscle Training on Foot Posture and Plantar Pressure Distribution in Individuals With Diabetic Foot Syndrome
Brief Title: Investigation of the Effect of Foot Intrinsic Muscle Training in Individuals With Diabetic Foot Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Fatma Dilara Akar, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-54
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; exercise; plantar pressure; intrinsic mucle training
MeSH Terms: conditions — Diabetic Foot; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1- Aerobic Exercise (Experimental): Group 1 participants will receive general foot care instructions and education on appropriate footwear selection, foot intrinsic muscle training, and in addition, an aerobic exercise protocol.
  Interventions: Other: Aerobic Exercise
- Group 2- Intrinsic Muscle Training (Experimental): Group 2 participants will receive general foot care instructions and education on appropriate footwear selection, along with an exercise protocol focusing on foot intrinsic muscle training.
  Interventions: Other: Intrinsic Muscle Training
- Group 3- Control Group (Experimental): Group 3 will receive only general foot care instructions and education on appropriate footwear selection.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — No intervention will be applied to the control group, and information will be given on general foot care instructions and the use of appropriate shoes.
  Arms: Group 3- Control Group
Other: Intrinsic Muscle Training — In addition to general foot care instructions and briefings on the use of appropriate shoes, intrinsic muscle training including alternating toe movement, toes picking up sheets, opening and closing the toes, pinching the toe separators, toe transitions and short foot exercises will be implemented.
  Additionaly, warm-up exercises, ankle exercises and functional exercises will be included in the program.
  Arms: Group 2- Intrinsic Muscle Training
Other: Aerobic Exercise — In addition to general foot care instructions and information on the use of appropriate shoes, warm-up exercises, ankle exercises, functional exercises and intrinsic muscle training, the participants will be given a walking program for aerobic exercise.
  Arms: Group 1- Aerobic Exercise

SUMMARY:
The goal of this experimental randomized controlled study is to evaluate the effectiveness of the exercise program to be applied to prevent foot wounds, which is one of the leading foot problems that develop as a result of diabetes, based on foot posture and plantar pressure distribution.

Participants who meet the inclusion criteria and are between the ages of 18-65 will be randomly assigned to one of the two experimental groups or the control group.Participants will be assessed through surveys to evaluate their physical activity level, foot health and functionality, and sensory status of the feet. Measurements related to foot position and posture will be taken. The use of a pedobarography device will allow for the examination of plantar pressure distribution. Following these assessments, participants will receive general foot care instructions and information on appropriate footwear, along with the designated exercise program.

During routine check-ups and treatment procedures related to diabetes, blood glucose levels and HbA1c values taken from participants will be analyzed by the physician before and after the program to make comparisons. The study is planned to last for 12 weeks, and evaluations will be conducted before and after the program.

DETAILED DESCRIPTION:
According to the literature, evaluations for preventing and treating diabetic foot ulcers commonly include plantar pressure measurements, and it is emphasized that methods involving plantar pressure technologies should be added to traditional evaluations to be more successful in preventing diabetic foot ulcers, even in high-risk individuals.

Based on the findings from previous research, it is believed that the reduced foot intrinsic muscle strength, which has not been extensively examined in its relationship with other factors, needs to be systematically investigated for its effects on foot related measurements and plantar pressure. Furthermore, there seems to be insufficient information regarding exercise interventions focusing on foot intrinsic muscle training for preventing ulcer development in diabetic foot. Therefore, the aim of the study is to examine the effects of foot intrinsic muscle training on foot posture and plantar pressure distribution in individuals with diabetic foot syndrome. By elucidating these factors, it is hoped that the exercise protocol focusing on foot intrinsic muscle training, implemented to prevent ulcer formation, will contribute to the literature and reduce the burdens associated with the disease.

Hypotheses of the study:

H0: Foot intrinsic muscle training has no effect on plantar pressure in individuals with diabetic foot syndrome.

H1: Foot intrinsic muscle training has an effect on plantar pressure in individuals with diabetic foot syndrome.

H2: Foot intrinsic muscle training has no effect on foot posture in individuals with diabetic foot syndrome.

H3: Foot intrinsic muscle training has an effect on foot posture in individuals with diabetic foot syndrome.

In this study, individuals with diabetic foot syndrome between the ages of 18-65 will be included. The study is designed as a randomized controlled trial, and the participants will be divided into three groups: one control group (Group 1) and two experimental groups (Group 2 and Group 3). The sample size was determined using the G-power program. According to the results obtained, it was calculated that a total of 30 individuals should be included in the study, with 10 participants in each group, considering a statistical power level of 82% and a significance level of 5%.

As part of the research, investigators will gain insights into participants' foot health through questionnaire questions, complete observational analyses of foot and foot-related measurements, evaluate participants' plantar pressure distribution using pedobarographic analysis, and implement exercise protocols focusing on foot intrinsic muscle training.

The study was designed with evaluation and treatment protocols. Demographic information and physical activity levels of the participants to be included in the study will be recorded. The measurements related to the foot will include evaluation of foot posture, goniometric measurements, assessment of tactile sensation, plantar pressure distribution analysis, and questionnaire evaluations. In addition to all these assessments, participants' blood values will be examined by the doctor before and after treatment.

The treatment protocols consist of general foot care instructions and information about appropriate footwear selection, along with exercise protocols. Group 1 - Control Group participants will receive only general foot care instructions and education on appropriate footwear selection. Group 2 participants will receive general foot care instructions and education on appropriate footwear selection, along with an exercise protocol focusing on foot intrinsic muscle training. Group 3 participants will receive general foot care instructions and education on appropriate footwear selection, foot intrinsic muscle training, and in addition, an aerobic exercise protocol. The treatment protocols will be implemented for 12 weeks, and pre- and post-treatment evaluations will be repeated to compare the results.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study voluntarily
* Be between the ages of 18-65
* Being diagnosed with type 1 or type 2 diabetes

Exclusion Criteria:

* Refusing to participate in the study or wanting to leave the study
* Presence of severe deformity and/or orthopedic problem in the foot
* Presence of foot ulcer
* History of lower extremity surgery
* History of lower extremity amputation
* Having serious comorbidities (renal failure, severe retinopathy, cardiac problems, neurological problems)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Plantar Pressure Distribution | 3 months
  Plantar pressure distribution analysis will be performed statically and dynamically with the Baropodometric Platforms Freemed™, 120 cm (Sensor Medica, Italia) pedobarography platform and software. In order to obtain the static plantar pressure distribution parameters of the people included in the study, on the surface with a pressure gauge sensor; As soon as the pressure falling on one foot reaches the value to be determined, it will be analyzed during standing static stance.

SECONDARY OUTCOMES:
Foot Posture | 3 months
  Foot Posture Index was used to evaluate the foot posture of the individuals to be included in the study. The assessment will be made by the therapist based on observation and palpation by asking individuals to stand still in a relaxed position where they feel comfortable. The talonavicular joint of the forefoot, medial longitudinal arch, and abduction/adduction of the forefoot relative to the hindfoot will be evaluated. In the hindfoot, eversion/inversion of the head of the talus, lateral malleolus, and calcaneus will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Akar, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the method and results of our study.
Supporting Information: Study Protocol
Time Frame: 3 months

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Morrison T, Jones S, Causby RS, Thoirs K. Can ultrasound measures of intrinsic foot muscles and plantar soft tissues predict future diabetes-related foot disease? A systematic review. PLoS One. 2018 Jun 15;13(6):e0199055. doi: 10.1371/journal.pone.0199055. eCollection 2018. PMID 29906277
- [Background] MANN R, INMAN VT. PHASIC ACTIVITY OF INTRINSIC MUSCLES OF THE FOOT. J Bone Joint Surg Am. 1964 Apr;46:469-81. No abstract available. PMID 14131426
- [Background] McKeon PO, Hertel J, Bramble D, Davis I. The foot core system: a new paradigm for understanding intrinsic foot muscle function. Br J Sports Med. 2015 Mar;49(5):290. doi: 10.1136/bjsports-2013-092690. Epub 2014 Mar 21. PMID 24659509
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Matos M, Mendes R, Silva AB, Sousa N. Physical activity and exercise on diabetic foot related outcomes: A systematic review. Diabetes Res Clin Pract. 2018 May;139:81-90. doi: 10.1016/j.diabres.2018.02.020. Epub 2018 Feb 23. PMID 29477503
- [Background] Lung CW, Wu FL, Liao F, Pu F, Fan Y, Jan YK. Emerging technologies for the prevention and management of diabetic foot ulcers. J Tissue Viability. 2020 May;29(2):61-68. doi: 10.1016/j.jtv.2020.03.003. Epub 2020 Mar 17. PMID 32197948
- [Background] Monteiro RL, Ferreira JSSP, Silva EQ, Donini A, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Feasibility and Preliminary Efficacy of a Foot-Ankle Exercise Program Aiming to Improve Foot-Ankle Functionality and Gait Biomechanics in People with Diabetic Neuropathy: A Randomized Controlled Trial. Sensors (Basel). 2020 Sep 9;20(18):5129. doi: 10.3390/s20185129. PMID 32916792
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Monteiro-Soares M, Russell D, Boyko EJ, Jeffcoate W, Mills JL, Morbach S, Game F; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the classification of diabetic foot ulcers (IWGDF 2019). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3273. doi: 10.1002/dmrr.3273. PMID 32176445
- [Background] Boulton AJ, Armstrong DG, Albert SF, Frykberg RG, Hellman R, Kirkman MS, Lavery LA, LeMaster JW, Mills JL Sr, Mueller MJ, Sheehan P, Wukich DK. Comprehensive foot examination and risk assessment. A report of the Task Force of the Foot Care Interest Group of the American Diabetes Association, with endorsement by the American Association of Clinical Endocrinologists. Phys Ther. 2008 Nov;88(11):1436-43. doi: 10.1093/ptj/88.11.1436. No abstract available. PMID 19137633
- See also: Feasibility of a home-based foot-ankle exercise programme for musculoskeletal dysfunctions in people with diabetes: randomised controlled FOotCAre (FOCA) Trial II. Sci Rep — https://doi.org/10.1038/s41598-021-91901-0